CLINICAL TRIAL: NCT00576849
Title: Phase 4 Study of a Total Balanced Volume Replacement Regimen in Elderly Cardiac Surgery Patients
Brief Title: A Total Balanced Volume Replacement Regimen in Elderly Cardiac Surgery Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Klinikum Ludwigshafen (Other)
Responsible Party: Prof. Dr. Joachim Boldt, Department of Anesthesiology and Intensive Care Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HES2007
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2009-01

CONDITIONS: Elderly; Cardiac Surgery
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Total balanced volume replacement regimen consisting of a balanced HES 130/0.42 plus a balanced crystalloid
  Interventions: Drug: Balanced HES 130/0.42
- B (Active Comparator): Conventional volume replacement strategy consisting of 6% HES 130/0.4 prepared in saline solution plus Ringer's lactate
  Interventions: Drug: 6% HES 130/0.4 prepared in saline solution

INTERVENTIONS:
Drug: Balanced HES 130/0.42 — Volume is administered perioperatively and during the first 48 hrs after surgery when mean arterial pressure (MAP) was <60mmHg and pulmonary capillary wedge pressure (PCWP) or central venous pressure (CVP) is <10 mmHg
  Arms: A
Drug: Balanced HES 130/0.42 — Volume will be administered perioperatively and during the first 48 hrs after surgery when mean arterial pressure (MAP) is <60mmHg and pulmonary capillary wedge pressure (PCWP) or central venous pressure (CVP) is <10 mmHg
  Arms: A
Drug: 6% HES 130/0.4 prepared in saline solution — Volume will be administered perioperatively and during the first 48 hrs after surgery when mean arterial pressure (MAP) is <60mmHg and pulmonary capillary wedge pressure (PCWP) or central venous pressure (CVP) is <10 mmHg
  Arms: B

SUMMARY:
A total balanced fluid replacement strategy is a promising concept for correcting hypovolemia. The effects of a balanced fluid management including a new balanced hydroxyethylstarch (HES) in elderly cardiac surgery patients will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >80 years

Exclusion Criteria:

* Chronic kidney dysfunction requiring dialysis
* Myocardial infarction within the previous 3 weeks
* Liver insufficiency

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is postoperative renal function | 28 days

SECONDARY OUTCOMES:
Other organ function (myocardial function, endothelial function, degree of inflammation) | Postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Boldt, M.D., Principal Investigator — Klinikum Ludwigshafen
Locations (1):
- Klinikum Ludwigshafen, Ludwigshafen, RLP, Germany